CLINICAL TRIAL: NCT02958618
Title: The Effect of Three Different Duration of Bolloon Dilation During ESBD in the Treatment of Common Bile Duct Stones
Brief Title: The Effect of Different Duration of Bolloon Dilation During ESBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PYZY16-011
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Common Bile Duct Stones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Duration for 30" group (Experimental): A limited sphincterotomy measuring up to one-third of the size of the papilla was first performed. Dilation with a controlled radial expansion (CRE) balloon (diameter 10, 12, 15, 18 ) was performed after the sphincterotomy. The balloon was centered at the sphincter and gradually filled with diluted contrast under endoscopic and fluoroscopic guidance until waisting was abolished. Once the waist had disappeared, the balloon was kept in position for 30 seconds. The stones were then removed by a basket or retrieval balloon. An ENBD catheter (.) was routinely placed into the CBD after stone removal.
  Interventions: Procedure: 30" group
- Duration for 60" group (Experimental): A limited sphincterotomy measuring up to one-third of the size of the papilla was first performed. Dilation with a controlled radial expansion (CRE) balloon (diameter 10, 12, 15, 18 ) was performed after the sphincterotomy. The balloon was centered at the sphincter and gradually filled with diluted contrast under endoscopic and fluoroscopic guidance until waisting was abolished. Once the waist had disappeared, the balloon was kept in position for 60 seconds. The stones were then removed by a basket or retrieval balloon. An ENBD catheter (.) was routinely placed into the CBD after stone removal.
  Interventions: Procedure: 60" group
- Duration for 180" group (Experimental): A limited sphincterotomy measuring up to one-third of the size of the papilla was first performed. Dilation with a controlled radial expansion (CRE) balloon (diameter 10, 12, 15, 18 ) was performed after the sphincterotomy. The balloon was centered at the sphincter and gradually filled with diluted contrast under endoscopic and fluoroscopic guidance until waisting was abolished. Once the waist had disappeared, the balloon was kept in position for 180 seconds. The stones were then removed by a basket or retrieval balloon. An ENBD catheter (.) was routinely placed into the CBD after stone removal.
  Interventions: Procedure: 180" group

INTERVENTIONS:
Procedure: 30" group — A limited sphincterotomy (EST) was performed prior to the EPBD.The length of the sphincterotomy incision was limited to a third of the size of the papilla. A CRE balloon (diameter 10, 12, 15, 18) was chosen according to the diameter of bile duct. The balloon was then gradually filled with diluted contrast medium under endoscopic and fluoroscopic guidance to observe the disappearance of the waist. Once the waist disappeared, the balloon remained inflated for 30 seconds. The stones were then retrieved by a basket or retrieval balloon. An ENBD catheter (.) was routinely placed into the CBD after stone removal.
  Arms: Duration for 30" group
Procedure: 60" group — A limited sphincterotomy (EST) was performed prior to the EPBD.The length of the sphincterotomy incision was limited to a third of the size of the papilla. A CRE balloon (diameter 10, 12, 15, 18) was chosen according to the diameter of bile duct. The balloon was then gradually filled with diluted contrast medium under endoscopic and fluoroscopic guidance to observe the disappearance of the waist. Once the waist disappeared, the balloon remained inflated for 60 seconds. The stones were then retrieved by a basket or retrieval balloon. An ENBD catheter (.) was routinely placed into the CBD after stone removal.
  Arms: Duration for 60" group
Procedure: 180" group — A limited sphincterotomy (EST) was performed prior to the EPBD.The length of the sphincterotomy incision was limited to a third of the size of the papilla. A CRE balloon (diameter 10, 12, 15, 18 ) was chosen according to the diameter of bile duct. The balloon was then gradually filled with diluted contrast medium under endoscopic and fluoroscopic guidance to observe the disappearance of the waist. Once the waist disappeared, the balloon remained inflated for 180 seconds. The stones were then retrieved by a basket or retrieval balloon. An ENBD catheter (.) was routinely placed into the CBD after stone removal.
  Arms: Duration for 180" group

SUMMARY:
Limited endoscopic sphincterotomy with balloon dilation（ESBD）is a promising technique in treating common bile duct stones. It had the similar success rate of stone extraction, but its incidence of complications remained uncertain. However, there is no clinical evidence and guideline to define the optimal duration of balloon dilation so far. So we designed a prospective randomized trial to compare the effect of three different duration of balloon dilation during ESBD so that we can find the optimal duration of the balloon dilation.

DETAILED DESCRIPTION:
Common Bile duct stones is one of the most common diseases of which the present incidence is 0.5% -3% in China. Endoscopic sphincterotomy (EST) is the most frequently used endoscopic technique for clearance of stones since the first description in 1974. Although EST is minimally invasive, it brings postoperative complications such as bleeding, perforation and acute pancreatitis. The overall complication and mortality is about 11.7-23% and 0.5%, respectively. Moreover, most believe EST can cause permanent sphincter of Oddi（SO） dysfunction which can result in biliary infection, stone recurrence and malignancies.

As an alternative method to EST, Endoscopic papillary balloon dilation (EPBD) was described by Staritz et al for the management of CBD stones. EPBD can preserve SO function and avoid undesirable effects due to an incompetent sphincter. It is reported that the basic SO function can be restored in one month after EPBD. Nonetheless, EPBD is indicated for the stones smaller than 12mm in diameters because the biliary orifice is enlarged to a lesser extent compared with EST. Furthermore, the incidence of postoperative pancreatitis reaches up to 15-30%. These disadvantages limit the application of EPBD.

As a result, Ersoz et al started a combined technique in 2003, which is called Endoscopic sphincterotomy with balloon dilation（ESBD）. ESBD can preserve SO function, reduce the adverse events, increase the stone removal rate. Especially, it can be applied for the stones larger than 12mm in diameters with large balloon dilatation. When ESBD is being performed, the duration of dilation is one of the most important factors affecting the postoperative complications. Whereas, there are issues regarding this technique that need further evaluation, such as the optimal duration of EPBD after EST. Some believe that short-term dilation can achieve the desired results and the duration of balloon dilation is not significantly correlated with postoperative pancreatitis, while opponents believe that although the small sphincterotomy is performed, short-term dilation has not been able to fully relax the residual sphincter. For long-term complications of ESBD, including the incidence of cholangitis, biliary stones recurrence rate, the incidence of biliary stenosis, there is no relative report either.

This prospective, randomized, controlled trial is designed to compare the difference of efficacy and morbidity among three different duration of balloon dilation（30s，60s，180s） after endoscopic sphincterotomy in the treatment of common bile duct stones. We hope that it will be helpful to establish the reasonable operation guidelines of ESBD.

ELIGIBILITY:
Inclusion Criteria:

* CBD stone patients, age≥18 years
* Stone diameter≤1.5cm

Exclusion Criteria:

* Unwilling to consent for the study
* Previous EST or EPBD
* Prior surgery of Bismuth Ⅱ and Roux-en-Y
* Benign or malignant CBD stricture
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease, primary sclerosing cholangitis (PSC), septic shock
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | Within 7 days after ESBD
  Patients with abdominal pain and serum amylase levels more than 3 times the upper limit of normal value. CT scanning is the best diagnostic discriminator

SECONDARY OUTCOMES:
Bleeding | Within 7 days after ESBD
  Haematemesis or malena is usually obvious immediately after sphincterotomy, but can be delayed for hours or even for several days.
Perforation | Within 7 days after ESBD
  Contrast or air is seen radiologically in the peritoneal cavity or the retroperitoneal region which can be routinely confirmed on CT
Acute cholangitis | Within 7 days after ESBD
  Patients typically present with fever, jaundice, and abdominal pain.
Pain | Within 7 days after ERCP
  Upper abdominal pain measured by Visual Analogue ScaleScore.
Success rate for clearance of stones | Within 72 hours after ERCP
  The success of stone removal is verified by the cholangiography after ESBD
Pancreatic duct insertion times | Within 24 hours after ESBD
  Times of the insertion of the duct or the guidewire into the pancreatic duct, no matter the depth
Operation time | Within 24 hours after ESBD
  From the insertion of the endoscope to the end of nasobiliary tube fixation
Hospital stay | Up to 30 days
  from the admission to the discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided